CLINICAL TRIAL: NCT06342167
Title: Efficacy and Safety of Concurrent Sintilimab and Radiotherapy With Immunonutrition Support in Esophageal Cancer: A Phase II Multicenter Clinical Trial
Brief Title: Efficacy and Safety of Concurrent PD-1 Inhibitor and Radiotherapy With Immunonutrition for Esophageal Squamous Cell Carcinoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, JIANYANG WANG, Principal Investigator, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC4409
Record Dates: First submitted 2024-03-26; First posted 2024-04-02 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Locally Advanced Esophageal Squamous Cell Carcinoma; Sintilimab; Radiotherapy; Concurrent Chemoradiotherapy; Immunonutrition
MeSH Terms: interventions — Radiotherapy; Immune Checkpoint Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Concurrent immunotherapy and radiotherapy (Experimental): Sintilimab + radiotherapy + enteral nutritional emulsion (TPF-T)
  Interventions: Radiation: Radiotherapy; Drug: Programmed Cell Death Protein 1 Inhibitor; Dietary Supplement: Immunonutrition support

INTERVENTIONS:
Radiation: Radiotherapy — Interventions consist of 50-60 Gy in 25-30 fractions of radiotherapy.
Drug: Programmed Cell Death Protein 1 Inhibitor — 200 mg of Sintilimab administered every three weeks concurrently with radiotherapy and after radiotherapy as consolidation therapy up to 1year.
  Other Names: PD-1 Inhibitor
Dietary Supplement: Immunonutrition support — 600-1600 ml of TPF-T per day according to the nutrition status evaluation
  Other Names: enteral nutritional emulsion

SUMMARY:
At present, concurrent chemoradiotherapy (cCRT) with platin-based dual-drug regimen is the standard treatment for inoperable, locally advanced esophageal cancer in patients with a good performance status. However, cCRT has substantial toxic effects, and a large number of patients with older age, malnutrition and other morbidities, cannot tolerate cCRT. Several phase II trials showed combining PD-1 inhibitor with definitive cCRT provided encouraging activity and acceptable toxicity in patients with locally advanced esophageal squamous cell carcinoma (LA-ESCC).

Therefore, this single-arm, multicenter, phase II trial aims to assess the efficacy and safety of immunotherapy plus radiotherapy with immunonutrition support in patients with LA-ESCC and positive PD-L1 expression who are intolerant to cCRT.

DETAILED DESCRIPTION:
This single-arm trial is designed to evaluate the efficacy and safety of concurrent immunotherapy (sintilimab) plus radiotherapy with immunonutrition support (enteral nutritional emulsion (TPF-T) followed by consolidation immunotherapy in inoperable patients with locally advanced or early stage esophageal squamous cell carcinoma , who are PD-L1 positive expression and intolerant to cCRT. The eligible patients will receive concurrent treatment consisting of total dose of 50-60 Gy in 25-30 fractions and 200 mg of sintilimab administered every three weeks, along with enteral nutritional emulsion (TPF-T) support (600-1600 ml per day according to the nutrition status evaluation). The primary outcome is 1-year progression-free survival (PFS) rate. The investigators hypothesized PD-L1 inhibitor plus radiotherapy will improve the 1-year PFS from 40% to 60%. Then, 58 patients will be needed in total. The secondary outcomes will include objective response rate (ORR), overall survival (OS), progression-free and overall survival, and incidence of adverse events.

This study is approval by the National GCP Center for Anticancer Drugs, Independent Ethics Committee, National Cancer Center/Cancer Hospital, Chinese Academy of Medical Science and Peking Union Medical College (Study ID: 24/074-4354).

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or order.
2. Diagnosed with locally advanced or early stage esophageal squamous cell carcinoma by pathological examinations of the primary lesion and imaging examinations, which are not resectable.
3. Confirmed to be unresectable and unable to tolerate synchronous chemoradiotherapy by multidisciplinary consultation, and has not undergone systemic drug therapy in the past.
4. PD-L1 tumor proportion score or combined positive score of ≥1%.
5. At least one measurable lesion on imaging according to the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
6. An Eastern Cooperative Oncology Group (ECOG) performance status score of 0 -2.
7. Expected survival time of more than three months.
8. Adequate organ function defined as the following laboratory indicators:

   1. Absolute neutrophil count (ANC) ≥ 1.5×109/L without use of granulocyte colony-stimulating factor in the past 14 days.
   2. Platelet count ≥ 100×109/L without blood transfusion in the past 14 days.
   3. Hemoglobin > 9g/dL without blood transfusion or use of erythropoietin-stimulating agents in the past 14 days.
   4. Total bilirubin ≤ 1.5×upper limit of normal (ULN).
   5. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5×ULN.
   6. Creatinine ≤ 1.5×ULN and creatinine clearance calculated using the Cockcroft-Gault formula) ≥ 60 ml/min.
   7. Good coagulation function, defined as an international normalized ratio (INR) or prothrombin time (PT) ≤ 1.5×ULN.
   8. Normal thyroid function, defined as thyroid-stimulating hormone (TSH) within the normal range. If the baseline TSH is outside the normal range, subjects with total T3 (or FT3) and FT4 within the normal range can still be included.
   9. Normal cardiac enzyme spectrum (or clinically insignificant laboratory abnormalities as determined by the investigator)
9. Negative pregnancy test (urine or serum) within 3 days before the first dose of study drug for female subjects of childbearing potential. If the urine pregnancy test cannot be confirmed as negative, a blood pregnancy test is required. Non-childbearing potential female is defined as postmenopausal for at least 1 year or has undergone surgical sterilization or hysterectomy.
10. Willing to sign the informed consent form.

Exclusion Criteria:

Subjects with any of the following conditions cannot participate in the study:

1. A high risk of bleeding or perforation due to clear invasion of adjacent organs (large arteries or trachea) by the tumor, or with fistula.
2. Diagnosed with malignancies other than esophageal cancer within 3 years prior to the first dose (excluding cured basal cell carcinoma or squamous cell carcinoma of the skin and/or radically resected carcinoma in situ).
3. Previous immunological or immunomodulatory drugs as systemic whole-body treatment, including thymic peptides, interferon, interleukins, except for local use to control pleural effusion.
4. Previous chest radiotherapy.
5. A history of allogeneic organ transplantation (except for corneal transplantation) or allogeneic hematopoietic stem cell transplantation.
6. Allergic to the study drug, Sintilimab, or its excipients.
7. A history of human immunodeficiency virus (HIV) infection (i.e., HIV1/2 antibody positive).
8. Untreated active hepatitis B defined as HBsAg positive and HBV-DNA copy number greater than the upper limit of the normal value in the laboratory of the study center.

   Note: Patients with hepatitis B who meet the following criteria can also be included:
   1. HBV viral load <1000 copies/ml (200IU/ml) before the first dose; the patient should receive anti-HBV treatment throughout chemotherapy in the entire study to avoid viral reactivation.
   2. For patients who are anti-HBc (+), HBsAg (-), anti-HBs (-), and HBV viral load (-), no prophylactic anti-HBV treatment is required, but close monitoring of viral reactivation is needed.
9. Active hepatitis C virus (HCV) infection defined as HCV antibody positive and HCV-RNA levels higher than the detection limit.
10. Having received live vaccines within 30 days prior to the first dose (Cycle 1, Day 1).

    Note: It is allowed to receive inactivated virus vaccines for seasonal influenza within 30 days prior to the first dose, but attenuated live influenza vaccines administered intranasally are not allowed.
11. Pregnant or lactating women;
12. Any serious or uncontrollable systemic diseases, such as:

    1. Significant and symptomatic abnormalities in rhythm, conduction or morphology on resting electrocardiogram, such as complete left bundle branch block, second-degree or higher heart block, ventricular arrhythmia, or atrial fibrillation;
    2. Unstable angina, congestive heart failure, or chronic heart failure classified as New York Heart Association (NYHA) class ≥ 2;
    3. Any arterial thrombosis, embolism or ischemic events, such as myocardial infarction, unstable angina, cerebrovascular accident or transient ischemic attack, occurring within 6 months prior to enrollment;
    4. Poor blood pressure control defined as systolic blood pressure > 140 mmHg and/or diastolic blood pressure > 90 mmHg;
    5. A history of non-infectious pneumonia requiring glucocorticoid therapy within 1 year prior to initial treatment, or current clinical activity of interstitial lung disease;
    6. Active pulmonary tuberculosis;
    7. Active or uncontrolled infections requiring systemic therapy;
    8. Active diverticulitis, abdominal abscess, or gastrointestinal obstruction;
    9. Liver diseases such as cirrhosis, decompensated liver disease, acute or chronic active hepatitis;
    10. Poorly controlled diabetes (fasting blood glucose (FBG) > 10mmol/L);
    11. Urine protein ≥ ++ on routine urinalysis, with confirmed 24-hour urine protein quantification > 1.0 g;
    12. Psychiatric disorders that are unable to comply with treatment.
13. Any other medical histories, disease evidence, treatment, or laboratory values that may interfere with the test results, hinder the full participation in the study, or other situations that the investigator deems unsuitable for inclusion due to potential risks.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Estimated)
Dates: Start 2024-03-14 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
1-year Progression-free survival rate (PFS) | From start of treatment until 1 years of follow-up.
  Progression-free survival rate is defined the rate of progress event at 1-years after radiotherapy. Progression event is defined as event of primary tumor and regional recurrence, or distant metastasis

SECONDARY OUTCOMES:
Objective response rate | Measured at 3 months after completion of radiotherapy
  Response is defined by the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
Progression-free survival | Measured at months 6, 12, 18, and 24.
  Progression-free survival is defined as the time from treatment to the event of primary tumor and regional recurrence, or distant metastasis
Overall survival rate | Measured at months 6, 12, 18, and 24.
  Live rate at months 6, 12, 18, and 24.
Overall survival | From start of treatment until 3 years of follow-up.
  Live status at different time points.
Incidence of adverse events | Measured at months 6, 12, 18, and 24.
  Adverse events are classified according to the Common Terminology Criteria for Adverse Events (CTCAE 5.0) criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Jianyang Wang, MD, Study Director — Cancer Institute and Hospital, Chinese Academy of Medical Sciences & Peking Union Medical College
Locations (9):
- China (9):
  - Department of Radiation Oncology, Cancer Institute and Hospital, Chinese Academy of Medical Sciences & Peking Union Medical College, Beijing, Beijing Municipality
  - Department of Radiation Oncology，Clinical Oncology School of Fujian Medical University，Fujian Cancer Hospital, Fujian, Fujian
  - Department of Oncology, Affiliated Hospital, Hebei University of Engineering, Handan, Hebei
  - Department 1st of Radiation Oncology, Anyang Tumor Hospital, Anyang, Henan
  - Department of Radiation Oncology the first affiliated hospital of Xinxiang Medical University, Xinxiang, Henan
  - Department of Radiation Oncology, General Hospital of Ningxia Medical University, Yinchuan, Ningxia
  - Department of Radiation Oncology，Fei County People's Hospital, Feixian, Shandong
  - Department of Radiation Oncology, Affiliated hospital of Jining Medical University, Jining, Shandong
  - Taizhou hospital of Wenzhou Medical University, Taizhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Park S, Oh D, Choi YL, Chi SA, Kim K, Ahn MJ, Sun JM. Durvalumab and tremelimumab with definitive chemoradiotherapy for locally advanced esophageal squamous cell carcinoma. Cancer. 2022 Jun 1;128(11):2148-2158. doi: 10.1002/cncr.34176. Epub 2022 Mar 23. PMID 35319779
- [Background] Zhu Y, Wen J, Li Q, Chen B, Zhao L, Liu S, Yang Y, Wang S, Lv Y, Li J, Zhang L, Hu Y, Liu M, Xi M. Toripalimab combined with definitive chemoradiotherapy in locally advanced oesophageal squamous cell carcinoma (EC-CRT-001): a single-arm, phase 2 trial. Lancet Oncol. 2023 Apr;24(4):371-382. doi: 10.1016/S1470-2045(23)00060-8. PMID 36990609
- [Background] Tachihara M, Tsujino K, Ishihara T, Hayashi H, Sato Y, Kurata T, Sugawara S, Shiraishi Y, Teraoka S, Azuma K, Daga H, Yamaguchi M, Kodaira T, Satouchi M, Shimokawa M, Yamamoto N, Nakagawa K; West Japan Oncology Group (WJOG). Durvalumab Plus Concurrent Radiotherapy for Treatment of Locally Advanced Non-Small Cell Lung Cancer: The DOLPHIN Phase 2 Nonrandomized Controlled Trial. JAMA Oncol. 2023 Nov 1;9(11):1505-1513. doi: 10.1001/jamaoncol.2023.3309. PMID 37676681
- [Background] Ohri N, Jolly S, Cooper BT, Kabarriti R, Bodner WR, Klein J, Guha C, Viswanathan S, Shum E, Sabari JK, Cheng H, Gucalp RA, Castellucci E, Qin A, Gadgeel SM, Halmos B. Selective Personalized RadioImmunotherapy for Locally Advanced Non-Small-Cell Lung Cancer Trial (SPRINT). J Clin Oncol. 2024 Feb 10;42(5):562-570. doi: 10.1200/JCO.23.00627. Epub 2023 Nov 21. PMID 37988638
- [Background] Li C, Tan L, Liu X, Wang X, Zhou Z, Chen D, Feng Q, Liang J, Lv J, Wang X, Bi N, Deng L, Wang W, Zhang T, Ni W, Chang X, Han W, Gao L, Wang S, Xiao Z. Concurrent chemoradiotherapy versus radiotherapy alone for patients with locally advanced esophageal squamous cell carcinoma in the era of intensity modulated radiotherapy: a propensity score-matched analysis. Thorac Cancer. 2021 Jun;12(12):1831-1840. doi: 10.1111/1759-7714.13971. Epub 2021 May 5. PMID 33949784
- [Background] Liu Y, Zheng Z, Li M, Zhang Y, Zhao F, Gong H, Lin H, Huang W, Chen X, Xu Z, Li X, Liu W, Cui Y, Zheng A, Li B. Comparison of concurrent chemoradiotherapy with radiotherapy alone for locally advanced esophageal squamous cell cancer in elderly patients: A randomized, multicenter, phase II clinical trial. Int J Cancer. 2022 Aug 15;151(4):607-615. doi: 10.1002/ijc.34030. Epub 2022 Apr 27. PMID 35419831
- [Background] Ji Y, Du X, Zhu W, Yang Y, Ma J, Zhang L, Li J, Tao H, Xia J, Yang H, Huang J, Bao Y, Du D, Liu D, Wang X, Li C, Yang X, Zeng M, Liu Z, Zheng W, Pu J, Chen J, Hu W, Li P, Wang J, Xu Y, Zheng X, Chen J, Wang W, Tao G, Cai J, Zhao J, Zhu J, Jiang M, Yan Y, Xu G, Bu S, Song B, Xie K, Huang S, Zheng Y, Sheng L, Lai X, Chen Y, Cheng L, Hu X, Ji W, Fang M, Kong Y, Yu X, Li H, Li R, Shi L, Shen W, Zhu C, Lv J, Huang R, He H, Chen M. Efficacy of Concurrent Chemoradiotherapy With S-1 vs Radiotherapy Alone for Older Patients With Esophageal Cancer: A Multicenter Randomized Phase 3 Clinical Trial. JAMA Oncol. 2021 Oct 1;7(10):1459-1466. doi: 10.1001/jamaoncol.2021.2705. PMID 34351356
- [Background] Chen Y, Ye J, Zhu Z, Zhao W, Zhou J, Wu C, Tang H, Fan M, Li L, Lin Q, Xia Y, Li Y, Li J, Jia H, Lu S, Zhang Z, Zhao K. Comparing Paclitaxel Plus Fluorouracil Versus Cisplatin Plus Fluorouracil in Chemoradiotherapy for Locally Advanced Esophageal Squamous Cell Cancer: A Randomized, Multicenter, Phase III Clinical Trial. J Clin Oncol. 2019 Jul 10;37(20):1695-1703. doi: 10.1200/JCO.18.02122. Epub 2019 Mar 28. PMID 30920880
- [Background] You J, Zhu S, Li J, Li J, Shen J, Zhao Y, Li X, Jia L, Li Q, Yang J, Wu Y, Shen W, Wu H, Wu X, Wang X, Ren Y, He J, Lin P, Zhu G, Shi A. High-Dose Versus Standard-Dose Intensity-Modulated Radiotherapy With Concurrent Paclitaxel Plus Carboplatin for Patients With Thoracic Esophageal Squamous Cell Carcinoma: A Randomized, Multicenter, Open-Label, Phase 3 Superiority Trial. Int J Radiat Oncol Biol Phys. 2023 Apr 1;115(5):1129-1137. doi: 10.1016/j.ijrobp.2022.11.006. Epub 2022 Nov 17. PMID 36402359
- [Derived] Yuan Y, Luo S, Wang X, Zheng Z, Qi Q, Wang Y, Chen M, Yang H, Gu P, Du Q, Wu X, Pan W, Xu Y, Wang J. Efficacy and safety of concurrent programmed cell death protein 1 inhibitor and definitive radiotherapy with immunonutrition support in esophageal squamous cell cancer: a phase II multicenter clinical trial. Radiat Oncol. 2025 Apr 18;20(1):58. doi: 10.1186/s13014-025-02604-z. PMID 40251674